CLINICAL TRIAL: NCT00097838
Title: A Phase I, Dose Escalation, Safety, and Immunogenicity Trial of an Alphavirus Replicon HIV-1 Subtype C Gag Vaccine (AVX101) in Healthy HIV-1 Uninfected Adult Participants
Brief Title: Safety of and Immune Response to an HIV-1 Subtype C Vaccine (AVX101) in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AlphaVax, Inc. (Industry)
Collaborators: HIV Vaccine Trials Network (Network); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 059
Record Dates: First submitted 2004-11-30; First posted 2004-12-01 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- 1 x 10^5 IU dose (Experimental): Vaccine dose of 1 x 10^5 IU per injection
  Interventions: Biological: AVX101
- 1 x 10^6 IU dose (Experimental): Vaccine dose of 1 x 10^6 IU per injection
  Interventions: Biological: AVX101
- 1 x 10^7 IU dose (Experimental): Vaccine dose of 1 x 10^7 IU per injection
  Interventions: Biological: AVX101
- 1 x 10^8 IU dose (Experimental): Vaccine dose of 1 x 10^8 IU per injection
  Interventions: Biological: AVX101
- Placebo (Placebo Comparator): phosphate buffered saline, pH 7.2, HSA, sodium gluconate, and sucrose
  Interventions: Other: placebo

INTERVENTIONS:
Biological: AVX101 — Alphavirus replicon particle vaccine expressing HIV Gag antigen
  Arms: 1 x 10^5 IU dose; 1 x 10^6 IU dose; 1 x 10^7 IU dose; 1 x 10^8 IU dose
Other: placebo — phosphate buffered saline, pH 7.2, HSA, sodium gluconate, and sucrose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of and immune response to an alphavirus replicon, HIV-1 subtype C gag vaccine, AVX101, in HIV uninfected adults in the United States, South Africa, and Botswana.

DETAILED DESCRIPTION:
HIV-1 subtype C is the prevailing subtype of HIV found in sub-Saharan Africa and is primarily responsible for the HIV/AIDS epidemic in southern Africa. Thus, development of a preventive subtype C vaccine is critically important in controlling the spread of HIV in this part of the world. This study will determine the safety and immunogenicity of an alphavirus replicon HIV-1 subtype C gag vaccine, AVX101, in HIV uninfected adults. This vaccine utilizes a propagation-defective replicon vector system derived from an attenuated strain of Venezuelan Equine Encephalitis (VEE) virus. The vaccine replicon expresses the gag gene from a South African subtype C isolate of HIV-1. Participants will be recruited in the United States, South Africa, and Botswana.

The study will last for 1 year. Participants will be enrolled sequentially, from lowest to highest dose of vaccine, into one of four groups. Groups will begin enrollment only following safety review of the previous group. Participants will be randomly assigned to receive active vaccine or placebo. During the study, participants will receive either 3 injections of one of four possible doses of the vaccine or 3 injections of placebo. Injections will be given at study entry and at Days 28 and 84. At screening, participants will undergo medical history assessment, a complete physical, HIV testing and counseling, and blood and urine collection; they will also be interviewed and asked to complete a questionnaire. After screening, there will be 8 study visits; the visits will occur at Days 14, 28, 42, 84, 98, 168, 273, and 364. Participants will be interviewed and asked to fill out a questionnaire at each study visit; participants will undergo a physical, additional HIV testing and counseling, and blood and urine collection at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* At low risk for HIV infection
* Willing to receive HIV test results
* Good general health
* Acceptable methods of contraception for females of reproductive potential
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus antibody (anti-HCV) negative or negative HCV PCR if anti-HCV is positive
* Meets educational requirements of the study

Exclusion Criteria:

* HIV vaccines or placebos in prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first study vaccine administration
* Blood products within 120 days prior to first study vaccine administration
* Immunoglobulin within 60 days prior to first study vaccine administration
* Live attenuated vaccines within 30 days prior to first study vaccine administration
* Investigational research agents within 30 days prior to first study vaccine administration
* Subunit or killed vaccines within 14 days prior to first study vaccine administration
* Allergy treatment with antigen injections within 30 days prior to first vaccine administration
* Current tuberculosis prophylaxis or therapy
* Serious adverse reaction to a vaccine. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Active syphilis
* Unstable asthma
* Type 1 or type 2 diabetes mellitus
* Thyroid disease requiring treatment in the past 12 months
* Serious angioedema within the past 3 years
* Uncontrolled hypertension
* Bleeding disorder
* Malignancy unless it has been surgically removed and, in the opinion of the investigator, is not likely to recur during the study period
* Seizure disorder requiring medication within the past 3 years
* Asplenia
* Mental illness that would interfere with compliance with the protocol
* Other conditions that, in the judgment of the investigator, would interfere with the study
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2004-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Grade IV adverse events | 1 year
  The sample size at each vaccine dose level was selected such that the stopping rule for not escalating the dose (2 or more vaccine-related Grade IV adverse experiences) would be met with high probability if the true toxicity rate was above 15-20%, and such that dose escalation would occur with high probability if the true toxicity rate was less than 5%.

SECONDARY OUTCOMES:
Local and systemic adverse events | 7 days after each dose
  Reactogenicity assessments were performed for all participants before and after each injection, beginning 25 to 45 minutes post injection and continuing daily for 7 days. Assessments performed included systemic reactogenicity (body temperature, malaise and/or fatigue, myalgia, headache, chills, arthralgia, nausea, vomiting) and local reactogenicity (injection site pain, tenderness, erythema or induration, and axillary lymph node tenderness or enlargement).
Binding antibodies by ELISA | 1 year
  Binding antibodies to commercially available Gag protein (P55 Gag; Quality Biologicals) were assessed by ELISA using single serum dilutions (1/50 or 1/100) on samples taken at baseline, two weeks after the second and third vaccinations and at the final visit. Samples that were positive in the initial ELISA were tested by endpoint titration ELISA using six 2- to 7-fold serial dilutions of serum beginning at a 1/50 or 1/100 dilution. Magnitude of responses is reported as the difference in optical density (OD) in antigen-containing and non-antigen containing wells at the 1:50 dilution.
Chromium release CTL assay | 3 months
  A standard 51Cr-release CTL assay was performed on fresh peripheral blood mononuclear cells (PBMC) at baseline and 2 weeks after the second and third vaccinations, using a 50:1 effector to target (E:T) ratio.
IFN-gamma ELISpot assay | 3 months
  Bulk T cell responses were assessed by IFN-γ ELISpot, using cryopreserved PBMC collected at baseline and 2 weeks after the second and third vaccinations, and stimulated overnight with Gag peptide pools at 200,000 cells per well.
Antibodies to VEE virus | 1 year
  Neutralizing antibodies to VEE virus were measured in serum obtained at baseline, 2 weeks after the second and third vaccinations and at the final visit.
Replication-competent viral vector viremia | 2 weeks after each vaccine dose
  Any participant who reported a fever greater than 38oC, or other moderate symptoms consistent with a viral illness (e.g. headache or malaise) during the 7 days following vaccination, or neurological symptoms (e.g. nuchal rigidity, ataxia, convulsions, coma, paralysis) within the window of the 2-week post vaccination visit, provided a serum sample to confirm the absence of replication-competent VEE viremia.
Intracellular cytokine staining (ICS) assay | 3 months
  Flow cytometry was used to examine HIV-specific CD4+ and CD8+ T cell responses using ICS, following stimulation with Gag peptides that span the protein sequence encoded by the vaccine construct. ICS assays were performed at baseline and 2 weeks after the second and third vaccinations.

CONTACTS AND LOCATIONS:
Overall Officials: Donald S. Burke, MD, Study Chair — Center for Immunization Research, Johns Hopkins School of Public Health; Salim Abdool Karim, MD, PhD, Study Chair — University of KwaZulu
Locations (8):
- United States (6):
  - Johns Hopkins University, Baltimore, Maryland
  - New York Blood Center - Union Square, New York, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - New York Blood Center - Bronx, The Bronx, New York
  - Vanderbilt University, Nashville, Tennessee
- Botswana HIV Vaccine Clinical Eval. Ctr, Princess, Gaborone, Botswana
- Perinatal HIV Research Unit, Chris Hani Baragwanat, Bertsham, South Africa

REFERENCES:
- [Background] Davis NL, West A, Reap E, MacDonald G, Collier M, Dryga S, Maughan M, Connell M, Walker C, McGrath K, Cecil C, Ping LH, Frelinger J, Olmsted R, Keith P, Swanstrom R, Williamson C, Johnson P, Montefiori D, Johnston RE. Alphavirus replicon particles as candidate HIV vaccines. IUBMB Life. 2002 Apr-May;53(4-5):209-11. doi: 10.1080/15216540212657. PMID 12120997
- [Background] Williamson AL. The development of HIV-1 subtype C vaccines for Southern Africa. IUBMB Life. 2002 Apr-May;53(4-5):207-8. doi: 10.1080/15216540212648. PMID 12120996
- [Background] Williamson C, Morris L, Maughan MF, Ping LH, Dryga SA, Thomas R, Reap EA, Cilliers T, van Harmelen J, Pascual A, Ramjee G, Gray G, Johnston R, Karim SA, Swanstrom R. Characterization and selection of HIV-1 subtype C isolates for use in vaccine development. AIDS Res Hum Retroviruses. 2003 Feb;19(2):133-44. doi: 10.1089/088922203762688649. PMID 12639249
- [Background] Schlesinger S. Alphavirus vectors: development and potential therapeutic applications. Expert Opin Biol Ther. 2001 Mar;1(2):177-91. doi: 10.1517/14712598.1.2.177. PMID 11727528
- [Derived] Wecker M, Gilbert P, Russell N, Hural J, Allen M, Pensiero M, Chulay J, Chiu YL, Abdool Karim SS, Burke DS; HVTN 040/059 Protocol Team; NIAID HIV Vaccine Trials Network. Phase I safety and immunogenicity evaluations of an alphavirus replicon HIV-1 subtype C gag vaccine in healthy HIV-1-uninfected adults. Clin Vaccine Immunol. 2012 Oct;19(10):1651-60. doi: 10.1128/CVI.00258-12. Epub 2012 Aug 22. PMID 22914365